CLINICAL TRIAL: NCT04464148
Title: Feasibility Trial of Pregnenolone for Posttraumatic Stress Disorder and Alcohol Use Disorder
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Feasibility study was not initiated.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sherwood Brown, MD, PhD, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU 2020-0171
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Post Traumatic Stress Disorder; Alcohol Use Disorder
Keywords: Pregnenolone; PTSD; Alcohol
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Pregnenolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pregnenolone 250 BID > Pregnenolone 400 BID (Experimental): For week 0-5 participants will receive pregnenolone 250 mg twice a day (total 500 mg/day). For weeks 6-8 participants will receive 400 mg twice a day (800 mg/day), if the drug is well tolerated.
  Interventions: Drug: Pregnenolone 250 mg; Drug: Pregnenolone 400 mg

INTERVENTIONS:
Drug: Pregnenolone 250 mg — Pregnenolone 250 mg capsule BID (500 mg QD total)
Drug: Pregnenolone 400 mg — Pregnenolone 400 mg capsule BID (800 mg QD total)

SUMMARY:
Pregnenolone is a neurosteroid and an over-the-counter supplement that has shown promise in clinical studies of stress-related disorders, such as anxiety, depression and posttraumatic stress disorder (PTSD). Epidemiological studies suggest that patients with PTSD are at higher risk of developing addiction, including alcohol use disorder (AUD).The following hypothesis will be tested in this trial: pregnenolone is associated with a reduction in both PTSD symptoms and the number of standard drinks per week in outpatients with PTSD and AUD.

DETAILED DESCRIPTION:
Investigators will conduct an 8-week, non-randomized, open label trial of pregnenolone in 20 persons with PTSD and AUD. The study will serve as a pilot study to determine feasibility and collect pilot data for NIH R01 proposals. All participants will be titrated to 800 mg/day of pregnenolone over the course of 4 weeks and maintain this dose for the remainder of the study. The study will consist of a screening visit to determine eligibility (Baseline I) and a Baseline II visit where participants will receive study medication, and follow-up visits at Weeks 1, 2, 3, 4, 6, and 8. Participants will complete a variety of assessments at each study visit, including clinician-rated and self-report measures of PTSD, alcohol use, depressive symptoms, cognitive performance, and side effects. Blood work will be done to ensure participant health and safety prior to randomization into the study, as well as to assess pregnenolone blood levels. All participants will meet with a study clinician at each visit to monitor safety and assess any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient adults (males and females) 18-70 years of age
* Meet criteria for current PTSD based on SCID-CV for DSM 5.
* Meet criteria for current AUD based on SCID-CV for DSM 5.
* Alcohol use of 14 standard drinks per week for men and 7 for women based on TLFB in the last week.
* Able to read and speak in English.
* If taking psychotropic medications, taking a stable dose for the past 2 weeks and during the study treatment.

Exclusion Criteria:

* Vulnerable populations (e.g., pregnancy/nursing, severe cognitive impairment, incarcerated).
* Current DSM-5 diagnosis of bipolar disorder, schizophrenia or other psychotic disorders based on SCID-CV.
* High risk for suicide (active SI with plan/intent or > 3 lifetime attempts in lifetime or any in the past 3 months).
* Coronary artery disease, atrial fibrillation, stroke, deep vein thrombosis, pulmonary embolism or blood clotting disorder, uncontrolled hypertension, cirrhosis or any severe, life threatening or unstable, medical condition as determined by clinician assessment.
* Clinically significant laboratory or physical examination findings.
* AST or ALT > 3 times the upper limit of normal.
* Evidence of clinically significant alcohol withdrawal symptoms defined as a CIWA-Ar score of ≥ 10.
* Current (last 14 days) treatment with naltrexone, acamprosate, disulfiram, topiramate.
* Intensive outpatient treatment (defined as ≥ 3 visits each week) for substance abuse (AA, NA meetings, or less intensive counseling at baseline will be allowed) or intensive psychosocial treatment for PTSD.
* Hormone-sensitive conditions (i.e. breast cancer; uterine/ovarian cancer, endometriosis, uterine fibroids).
* Use of oral contraceptives or hormone replacement therapy.
* History of allergic reaction or side effects with prior pregnenolone use.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Baseline to 8 weeks
  CAPS-5 is a 30-item questionnaire, corresponding to the DSM-5 diagnosis for PTSD. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms. Similarly, CAPS-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms corresponding to a given DSM-5 cluster: Criterion B (items 1-5); Criterion C (items 6-7); Criterion D (items 8-14); and, Criterion E (items 15-20). A symptom cluster score may also be calculated for dissociation by summing items 19 and 20. The higher scores are associated with greater PTSD severity.
Standard alcoholic drinks per week | Baseline to 8 weeks
  The Timeline Followback will be used to assess the change in the number of standard alcoholic drinks per week. The TLFB will be administered by an interviewer and involves asking participants to retrospectively estimate their alcohol use 28 days prior to the first appointment and between each visit. The reported drinks are then converted to standard drinks based on the drink's alcohol by volume (ABV). The higher number is associated with more standard drinks and worse outcome.
Timeline Followback (TLFB) heavy drinking days | Baseline to 8 weeks
  The Timeline Followback will be used to assess the change in the number of standard alcoholic drinks per week. The TLFB will be administered by an interviewer and involves asking participants to retrospectively estimate their alcohol use 28 days prior to the first appointment and between each visit. The reported drinks are then converted to heavy drinking days based on the drink's alcohol by volume (ABV) and participant's sex (male/female) - 5 drinks per day for males and 4 for females. Each day during which 4-5 drinks are consumed is counted as a heavy drinking day within a given assessment period. The higher number is associated with more heavy drinking days and worse outcome.
Systematic Assessment for Treatment Emergent Events (SAFTEE) | Baseline to 8 weeks
  SAFTEE is a side effect self-report assessment scale that consists of 56 potential side effects. Participants rate how bothersome each side effect is on a scale of "none" (0), "mild" (1), "moderate" (2), "severe" (3). The higher total score (all items summed together) indicates a higher level of side effect burden.
Patient-rated PTSD Checklist for DSM-5 (PCL-5). | Baseline to 8 weeks
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The self-report rating scale is 0-4 for each symptom, reflecting a change from 1-5 in the DSM-IV version. Rating scale descriptors correspond to "Not at all" (0), "A little bit" (1), "Moderately" (2), "Quite a bit" (3), and "Extremely" (4).A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. The higher score is associated with poorer outcome.

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, MD, PhD, MBA, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No